CLINICAL TRIAL: NCT05380973
Title: Clinical Evaluation of Two Fiber Reinforced Resin Composites Versus Nanohybrid Resin Composite in Posterior Restorations: Randomized Clinical Trial
Brief Title: Clinical Performance of Two Fiber Reinforced Resin Composites Versus Nanohybrid Resin Composite in Posterior Teeth Will be Evaluated Using Modified USPHS Criteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Mohamed Kamal, Assistant lecturer, conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fiber reinforced composite
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Dental Restoration Failure
Keywords: polyethylene fiber reinforced resin composite; glass fiber reinforced resin composite; nanohybrid resin composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fiber reinforced resin composite (Experimental): Short fiber resin composite (SFRC) (Ever X Posterior, GC, Japan) The material will be applied according to manufacturer instructions. A thin layer of flowable resin composite will be applied prior placing the short fiber reinforced composite, then SFRC (Ever X Posterior, GC, Tokyo, Japan) will be injected in bulk, and light cured for 20 seconds, nanohybrid resin composite will be placed to the rest of the cavity incrementally.
  Polyethylene ribbon fiber (Ribbond Inc., Seattle, WA, USA) The material will be applied according to manufacturer instructions. After application of a thin layer of the flowable resin composite to the cavity, a layer of Polyethylene ribbon fiber on the unpolymerized flowable composite will be condensed with a plugger and polymerized for 20 seconds then, nanohybrid resin composite will be placed to the rest of the cavity incrementally.
  Interventions: Other: Short fiber resin composite; Other: Polyethylene ribbon fiber
- Nanohybrid resin composite (Active Comparator): A thin layer of flowable composite will be applied then nanohybrid resin composite will be applied to the rest of the cavity using the conventional incremental technique according to manufacturer instructions.
  Interventions: Other: Short fiber resin composite; Other: Polyethylene ribbon fiber

INTERVENTIONS:
Other: Short fiber resin composite — resin composite reinforced with short glass fibers
  Other Names: (Ever X Posterior, GC, Japan)
Other: Polyethylene ribbon fiber — resin composite reinforced with polyethylene ribbon fiber
  Other Names: (Ribbond Inc., Seattle, WA, USA)

SUMMARY:
This study is conducted to evaluate the clinical performance of two fiber-reinforced resin composite restorations compared to nanohybrid resin composite restorations in patients with posterior MOD cavities

DETAILED DESCRIPTION:
Statement of the problem:

With limited evidence based information in literature about using fiber-reinforced composite (FRC) restorations in stress bearing posterior areas, it is beneficial to evaluate the newly introduced materials using a randomized clinical trial to test the null hypothesis that this new material "fiber reinforced resin composites" will have the same clinical performance as the nanohybrid resin composite restoration in such situation

Rationale:

Improvements concerning the esthetic and mechanical properties of dental resin composites have resulted in widespread use of these materials in both anterior and posterior teeth. However, resin composites still have a number of limitations in posterior teeth, mainly because of problems related to technique sensitivity, polymerization shrinkage and low fracture resistance, Due the failures of this kind, it is still controversial, whether restorative composites should be used in large high-stress bearing applications such as in direct posterior restorations.

Fiber-reinforcement of resin-based composite restorations has been proposed to increase resistance of materials fracturing under high stress-bearing cavities. Fiber-reinforced composite (FRC) is made of a polymer matrix, impregnated with fibers. The fibers allow the stresses to be distributed throughout the restoration. Since the role of the fibers is to improve the structura lproperties of the material by acting as crack stoppers, the FRC framework provides strength and rigidity of the composite materials.

The common types of fibers used in dentistry are glass and polyethylene fibers. Composite resin reinforced with short E-glass fiber fillers showed substantial improvements in the load bearing capacity, the flexural strength and fracture toughness of in comparison with conventional particulate filler restorative composite resin. The short fiber composite resin has also revealed control of the polymerization shrinkage stress by fiber orientation and, thus, marginal microleakage was reduced compared with conventional particulate filler restorative composite resins.

Polyethylene fibers are one of the most durable reinforcing fibers available. They are made of aligned polymer chains, having low modulus and density, and presents good impact resistance.They are white in colour and thus it is possible to use them in aesthetic dental applications, the use of polyethylene fiber ribbon in combination with bonding agent and flowable composite under composite restoration may act as a stress absorber because of its lower elastic modulus thereby increasing fracture resistance

ELIGIBILITY:
Inclusion Criteria:

* MOD carious lesions premolars and molars.
* Vital upper or lower teeth with no signs of irreversible pulpitis.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Deep carious defects (close to pulp, less than 1 mm distance).
* Periapical pathology or signs of pulpal pathology.
* Endodontically treated teeth.
* Tooth hypersensitivity.
* Possible prosthodontic restoration of teeth.
* Heavy occlusion and occlusal contacts or history of bruxism
* Severe periodontal affection.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Change in the clinical performance | Change from the baseline at 12 months.
  Measured using modified USPHS criteria for clinical evaluation of restoration failure.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Sayed Mosallam, Study Director — Professor
Locations (1):
- faculty of dentistry-Cairo university, Cairo, Egypt

REFERENCES:
- [Derived] Mohamed MH, Abouauf EA, Mosallam RS. Clinical performance of class II MOD fiber reinforced resin composite restorations: an 18-month randomized controlled clinical trial. BMC Oral Health. 2025 Jan 30;25(1):159. doi: 10.1186/s12903-025-05521-5. PMID 39881262